CLINICAL TRIAL: NCT05991596
Title: Vitiligo and Psychological Distress: Pilot Study for the Experimentation of a Psychodramatic Psychotherapy Treatment
Brief Title: Vitiligo and Psychodrama Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Provinciale per i Servizi Sanitari, Provincia Autonoma di Trento (Other)
Collaborators: Università degli Studi di Brescia (Other); Scuola Psicoterapia Psicodrammatica Brescia (Unknown); Università degli Studi di Trento (Other)
Responsible Party: Principal Investigator, Gabriella Pravata, Medical Doctor, Dermatologist, Azienda Provinciale per i Servizi Sanitari, Provincia Autonoma di Trento
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A800
Record Dates: First submitted 2023-07-26; First posted 2023-08-14 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychodramatic Psychotherapy (Experimental): This experimental arm will include 12 patients with vitiligo (randomly assigned to this arm), attending the dermatology services of APSS Trento.
  This experimental group will receive the drug treatment usually recommended for vitiligo, in addition to 6 months of psychodramatic psychotherapy.
  Interventions: Behavioral: Psychodramatic psychotherapy
- Self-help activities (Active Comparator): This is a control arm which will include 12 patients with vitiligo (randomly assigned to this arm), attending the dermatology services of APSS Trento. This control group will receive the drug treatment usually recommended for vitiligo, in addition to 6 months of self-help activities.
  Interventions: Behavioral: Self-help activities

INTERVENTIONS:
Behavioral: Psychodramatic psychotherapy — The psychodramatic psychotherapy will include a total of 14 meetings during a 6 months period and they will be held in presence (or remotely in case of COVID-19 government restrictions) as follows:
  * 1 individual motivational interview;
  * 1 weekly group session lasting 2 hours for 1 month (total 4 meetings);
  * 1 group session every 15 days lasting 2 hours, for 5 months (total 10 meetings).
  Patients will also receive the pharmacological treatment usually recommended for vitiligo.
  Arms: Psychodramatic Psychotherapy
Behavioral: Self-help activities — The self-help activities will include:
  * 1 individual motivational interview;
  * 1 weekly, 2 hours group meeting, for 1 month (total 4 meetings);
  * 1 group meeting lasting 2 hours every 15 days, for 5 months (total 10 meetings).
  Patients will also receive pharmacological treatment usually recommended for vitiligo.
  Arms: Self-help activities

SUMMARY:
The goal of this pilot clinical trial is to assess the effectiveness of psychodramatic psychotherapy in reducing the psychological distress and/or the skin condition in patients with vitiligo.

The main questions it aims to answer are:

1. Is there any improvement in terms of psychological distress in patients with vitiligo participating in a psychodramatic psychotherapy, compared to a control group?
2. Is there any improvement in terms of skin condition in patients with vitiligo participating in a psychodramatic psychotherapy, compared to a control group? Participants in the experimental group will receive the dermatological drug treatment usually recommended for vitiligo, and in addition they will participate in a 6 months psychodramatic psychotherapy.

Researchers will compare the results of the experimental group with the results of a control group including vitiligo patients who will receive the dermatological pharmacological treatment usually recommended for vitiligo and participate in a 6 months program of self-help activities.

DETAILED DESCRIPTION:
The primary aim of this pilot study is to assess any possible improvement in terms of psychological distress in patients with vitiligo participating in a psychodramatic psychotherapy (PSD), in addition to the usual pharmacological treatment with hydrocortisone and heliotherapy.

The secondary aim is to assess any improvement in terms of vitiligo skin condition and/or other systemic autoimmune diseases symptoms.

The study will involve 24 patients with vitiligo aged between 18 and 55 years, attending the dermatology services of the Azienda Provinciale per i Servizi Sanitari (APSS) of Trento.

Patients will be randomly assigned to one of the two groups:

* 12 patients will receive the dermatological pharmacological treatment usually recommended for vitiligo, and in addition they will participate in a psychodramatic group psychotherapy for 6 months (PSD experimental group);
* 12 patients will receive the dermatological pharmacological treatment usually recommended for vitiligo, and in addition they will receive self-help activities for 6 months (non-PSD control group).

The experimental group (PSD) will attend the psychodramatic psychotherapy, which will include:

* 1 individual motivational interview;
* 1 weekly group session lasting 2 hours for 1 month (total 4 meetings);
* 1 group session every 15 days lasting 2 hours, for 5 months (total 10 meetings).

The control group (non-PSD) will attend self-help activities as follows:

* 1 individual motivational interview;
* 1 weekly, 2 hours group meeting, for 1 month (total 4 meetings);
* 1 group meeting lasting 2 hours every 15 days, for 5 months (total 10 meetings).

To all patients participating in the study, the following pharmacological treatment will be administered:

* Hydrocortisone acetate with the following dosage: 1 Finger Unit /15 cm2 per day. Duration: 10 days a month for 6 months.
* Free exposure to the sun without photoprotection from 9.00 AM to 11.00 AM.

A clinical evaluation will be carried out at:

Time 0 (T0): right before the beginning of the intervention Time 1 (T1): after 6 months, at the end of the intervention For both groups, a follow-up will be performed after 6 months from the end of the intervention (psychodramatic psychotherapy or self-help activities).

ELIGIBILITY:
Inclusion Criteria:

1. Segmental vitiligo with unilateral localization.
2. Non-segmental vitiligo (acrofacial; mucosal with more than one side affected; generalized universal; mixed associated with segmental vitiligo).
3. Vitiligo-associated autoimmune comorbidity referred to in points 1-2: Thyroiditis.
4. Symptoms of depression and/or anxiety and/or low self-esteem associated with Vitiligo mentioned in points 1-2.

Exclusion Criteria:

* Cognitive impairment/dementia (clinically diagnosed).
* Individual and/or group psychotherapy in progress.
* Have previously received other psychotherapy.
* Use of psychiatric drugs in the last 3 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2023-11-02 (Actual); Primary Completion 2024-05-11 (Actual); Study Completion 2024-05-11 (Actual)

PRIMARY OUTCOMES:
Improvement of the levels of psychological distress of patients with vitiligo | Time 0: Before the beginning of the intervention; Time 1: after 6 months, at the end of the intervention
  The General Health Questionnaire (GHQ-12), a self-administered questionnaire covering several domains associated with a person's psychological well-being, will be administered to all patients. Scoring is along a 4-point scale (total score ranging from 0 to 36) with higher scores suggestive of more distress.
Improvement of the levels of psychological distress of patients with vitiligo, in terms of psychological, functional or physical state. | Time 0: Before the beginning of the intervention; Time 1: after 6 months, at the end of the intervention
  The Short-Form Health Survey (SF-36): a health status profile originally designed to measure health status and outcomes, will be administered to all patients. This instrument addresses health concepts from the patient's perspective and its 36 questions are meant to reflect 8 domains of health, evaluating any changes in the psychological, functional or physical state of patients. SF-36 scores range from 0 (worst) to 100 (best).
Improvement of the levels of psychological distress of patients with vitiligo, in terms of anxiety symptoms | Time 0: Before the beginning of the intervention; Time 1: after 6 months, at the end of the intervention
  The Beck Anxiety Inventory (B.A.I.), a self-report measure of anxiety, will be administered to all patients. The BAI items are scored on a scale between 0 and 3 and have a maximum score of 63, with higher scores suggestive of higher levels of anxiety.
Improvement of the levels of psychological distress of patients with vitiligo, in terms of depressive symptoms | Time 0: Before the beginning of the intervention; Time 1: after 6 months, at the end of the intervention
  The Beck Depression Inventory (B.D.I.), a 21-question multiple-choice self-report inventory and one of the most widely used instruments for measuring the severity of depression, will be administered to all patients. A value of 0 to 3 is assigned for each answer and then the total score is compared to a key to determine the depression's severity. Higher total scores indicate more severe depressive symptoms.
Improvement of the levels of psychological distress of patients with vitiligo, in terms of spontaneity | Time 0: Before the beginning of the intervention; Time 1: after 6 months, at the end of the intervention
  The Revised Spontaneity Assessment Inventory (SAI-R) will be administered to all patients. The SAI-R is a scale for the assessment of spontaneity, evaluating feelings and thoughts that people experience in different daily situations. It includes 18 items, scored on a 5-point Likert scale. Higher total scores indicate higher levels of spontaneity (score range: 18-90)

SECONDARY OUTCOMES:
Improvement of vitiligo and/or other systemic autoimmune diseases symptoms, in terms of dermatological lesions related to vitiligo and any re-pigmentation | Time 0: Before the beginning of the intervention; Time 1: after 6 months, at the end of the intervention
  The Vitiligo Extent Score (VES) will be administered. The VES will be administered at Time 0 in order to evaluating the extent of vitiligo, and at Time 1 to evaluate any repigmentation. The VES is a template of vitiligo images that measures vitiligo at 19 different areas of the body. The physician has to score these 19 body areas separately by selecting the image that most resembles to patient's clinical in that body area, ranging from no lesion to almost 100% lesion coverage.
Improvement of vitiligo and/or other systemic autoimmune diseases symptoms, in terms of personal perception of the patient | Time 0: Before the beginning of the intervention; Time 1: after 6 months, at the end of the intervention
  The Self Administered version of Vitiligo Extent score (SA-VES) will be administered. The SA-VES is a patient-reported outcome measurement instrument that is similar to the VES (it includes only 12 areas). It will be self- administered at Time 0 in order to evaluating the extent of vitiligo, and at Time 1 to evaluate any repigmentation.
Improvement of vitiligo and/or other systemic autoimmune diseases symptoms, in terms of quality of life associated with the skin condition | Time 0: Before the beginning of the intervention; Time 1: after 6 months, at the end of the intervention
  Skindex-29, a three-dimensional, dermatology-specific Health-related quality of life questionnaire, will be administered. Skindex-29 items are combined to form three domains: symptoms, emotions, and functioning. The domain scores and an overall score are expressed on a 100-point scale, with higher scores indicating lower levels of quality of life.
Multidimensional improvement of vitiligo | Time 0: Before the beginning of the intervention; Time 1: after 6 months, at the end of the intervention
  An adaptation of the Vitiligo Questionnaire ITA 4.0 will be administered. The Vitiligo Questionnaire ITA 4.0 measures several aspects of health status in vitiligo patients. It is self-administered and features thirty questions in five sections. These cover biologic factors, symptom status, functional status, treatment outcome perception, and economic impact.
Improvement of other autoimmune diseases, in terms of levels of levels of Thyroid Stimulating Hormone | Time 0: Before the beginning of the intervention; Time 1: after 6 months, at the end of the intervention
  Blood chemistry tests will be conducted to assess levels of Thyroid Stimulating Hormone (TSH), a pituitary thyroid-stimulating hormone that regulates thyroid activity. Reference values are 0.2-4.5 mU/L. Higher values may indicate thyroid hormone deficiency, lower levels may indicate thyroid hormone excess.
Improvement of other autoimmune diseases, in terms of levels of S-Free T4-Thyroxine | Time 0: Before the beginning of the intervention; Time 1: after 6 months, at the end of the intervention
  Blood chemistry tests will be conducted to assess levels of S-Free T4-Thyroxine (FT4), a thyroid hormone that regulates the body's metabolism, secretion of which is controlled by thyroid-stimulating hormone (TSH) produced by the pituitary gland. Reference values are 12.0 - 22.0 pmol/L. Higher values may indicate hyperthyroidism, lower levels may indicate hypothyroidism.
Improvement of other autoimmune diseases, in terms of levels of Anti Thyroglobulin | Time 0: Before the beginning of the intervention; Time 1: after 6 months, at the end of the intervention
  Blood chemistry tests will be conducted to assess levels of Anti Thyroglobulin (HTG), antibodies produced against thyroglobulin, a precursor protein of thyroid hormones triiodothyronine (FT3) and free thyroxine (FT4), indicating autoimmune pathology. Threshold value is 115 IU/ml; higher values may indicate possible development of hypothyroidism.
Improvement of other autoimmune diseases, in terms of levels of Anti Thyroperoxidase | Time 0: Before the beginning of the intervention; Time 1: after 6 months, at the end of the intervention
  Blood chemistry tests will be conducted to assess levels of Anti Thyroperoxidase (TPO), an antibody which, attacking the enzyme peroxidase, identifying autoimmune thyroid disease.
  Threshold value is 34 IU/ml; higher values may be associated with either hyperthyroidism or hypothyroidism (depending on whether it's Graves' disease or Hashimoto's thyroiditis).
Improvement of other autoimmune diseases, in terms of levels of Antinuclear Antibodies | Time 0: Before the beginning of the intervention; Time 1: after 6 months, at the end of the intervention
  Blood chemistry tests will be conducted to assess levels of Antinuclear Antibodies (ANA), antibodies produced by the body's immune system, indicating the presence of autoantibodies in circulating blood.
  Threshold value is 1:160.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Pravatà, MD, Principal Investigator — APSS Trento
Locations (1):
- APSS Trento, Trento, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bassi R. Psiche e pelle. Introduzione alla dermatologia psicosomatica. 2006; Ed. Bollati Boringheri, Torino.
- [Background] Bottaccioli F, Bottaccioli MG. Psiconeuroendocrinoimmunologia e scienza della cura integrata (pp 197-203; 203-210). 2017; Ed. Edra.
- [Background] Bottaccioli F. Epigenetica e PNEI. 2016; Ed. Edra.
- [Background] Arck PC, Slominski A, Theoharides TC, Peters EM, Paus R. Neuroimmunology of stress: skin takes center stage. J Invest Dermatol. 2006 Aug;126(8):1697-704. doi: 10.1038/sj.jid.5700104. PMID 16845409
- [Background] Chapman BP, Moynihan J. The brain-skin connection: role of psychosocial factors and neuropeptides in psoriasis. Expert Rev Clin Immunol. 2009 Nov;5(6):623-7. doi: 10.1586/eci.09.56. No abstract available. PMID 20477685
- [Background] Alhetheli GI. The Impact of Vitiligo on Patients' Psychological Status and Sexual Function: Cross-Sectional Questionnaire-Based Study. The Open Dermatology Journal. 2021; 15: 23-30.
- [Background] Taneja K, Taneja J, Kaur C, Patel S, Haldar D. Lipid Risk Factors in Vitiligo: Homocysteine the Connecting Link? Clin Lab. 2020 Oct 1;66(10). doi: 10.7754/Clin.Lab.2020.200120. PMID 33073941
- [Background] Hamzavi I, Jain H, McLean D, Shapiro J, Zeng H, Lui H. Parametric modeling of narrowband UV-B phototherapy for vitiligo using a novel quantitative tool: the Vitiligo Area Scoring Index. Arch Dermatol. 2004 Jun;140(6):677-83. doi: 10.1001/archderm.140.6.677. PMID 15210457
- [Background] Papadopoulos L, Bor R, Legg C, Hawk JL. Impact of life events on the onset of vitiligo in adults: preliminary evidence for a psychological dimension in aetiology. Clin Exp Dermatol. 1998 Nov;23(6):243-8. doi: 10.1046/j.1365-2230.1998.00384.x. PMID 10233617
- [Background] Picardi A, Pasquini P, Cattaruzza MS, Gaetano P, Melchi CF, Baliva G, Camaioni D, Tiago A, Abeni D, Biondi M. Stressful life events, social support, attachment security and alexithymia in vitiligo. A case-control study. Psychother Psychosom. 2003 May-Jun;72(3):150-8. doi: 10.1159/000069731. PMID 12707482
- [Background] Ongenae K, Beelaert L, van Geel N, Naeyaert JM. Psychosocial effects of vitiligo. J Eur Acad Dermatol Venereol. 2006 Jan;20(1):1-8. doi: 10.1111/j.1468-3083.2005.01369.x. PMID 16405601
- [Background] Porter J, Beuf A, Nordlund JJ, Lerner AB. Personal responses of patients to vitiligo: the importance of the patient-physician interaction. Arch Dermatol. 1978 Sep;114(9):1384-5. No abstract available. PMID 686757
- [Background] Porter J, Beuf AH, Nordlund JJ, Lerner AB. Psychological reaction to chronic skin disorders: a study of patients with vitiligo. Gen Hosp Psychiatry. 1979 Apr;1(1):73-7. doi: 10.1016/0163-8343(79)90081-1. PMID 499777
- [Background] Ezzedine K, Silverberg N. A Practical Approach to the Diagnosis and Treatment of Vitiligo in Children. Pediatrics. 2016 Jul;138(1):e20154126. doi: 10.1542/peds.2015-4126. Epub 2016 Jun 21. PMID 27328922
- [Background] Shenefelt PD. Mindfulness-Based Cognitive Hypnotherapy and Skin Disorders. Am J Clin Hypn. 2018 Jul;61(1):34-44. doi: 10.1080/00029157.2017.1419457. PMID 29771216
- [Background] Shah R, Hunt J, Webb TL, Thompson AR. Starting to develop self-help for social anxiety associated with vitiligo: using clinical significance to measure the potential effectiveness of enhanced psychological self-help. Br J Dermatol. 2014 Aug;171(2):332-7. doi: 10.1111/bjd.12990. Epub 2014 Aug 4. PMID 24665869
- [Background] Papadopoulos L, Bor R, Legg C. Coping with the disfiguring effects of vitiligo: a preliminary investigation into the effects of cognitive-behavioural therapy. Br J Med Psychol. 1999 Sep;72(3):385-96. doi: 10.1348/000711299160077. PMID 10524722
- [Background] Picardi A, Abeni D, Melchi CF, Puddu P, Pasquini P. Psychiatric morbidity in dermatological outpatients: an issue to be recognized. Br J Dermatol. 2000 Nov;143(5):983-91. doi: 10.1046/j.1365-2133.2000.03831.x. PMID 11069507
- [Background] Osinubi O, Grainge MJ, Hong L, Ahmed A, Batchelor JM, Grindlay D, Thompson AR, Ratib S. The prevalence of psychological comorbidity in people with vitiligo: a systematic review and meta-analysis. Br J Dermatol. 2018 Apr;178(4):863-878. doi: 10.1111/bjd.16049. Epub 2018 Feb 7. PMID 28991357
- [Background] Ramakrishna P, Rajni T. Psychiatric morbidity and quality of life in vitiligo patients. Indian J Psychol Med. 2014 Jul;36(3):302-3. doi: 10.4103/0253-7176.135385. PMID 25035556
- [Background] Simons RE, Zevy DL, Jafferany M. Psychodermatology of vitiligo: Psychological impact and consequences. Dermatol Ther. 2020 May;33(3):e13418. doi: 10.1111/dth.13418. Epub 2020 May 4. PMID 32297399
- [Background] Cupertino F, Niemeyer-Corbellini JP, Ramos-E-Silva M. Psychosomatic aspects of vitiligo. Clin Dermatol. 2017 May-Jun;35(3):292-297. doi: 10.1016/j.clindermatol.2017.01.001. Epub 2017 Jan 21. PMID 28511827
- [Background] Moreno JL. Manuale di Psicodramma Vol. I e Vol. II. 1987; Ed. Astrolabio
- [Background] Orkibi H, Feniger-Schaal R. Integrative systematic review of psychodrama psychotherapy research: Trends and methodological implications. PLoS One. 2019 Feb 19;14(2):e0212575. doi: 10.1371/journal.pone.0212575. eCollection 2019. PMID 30779787
- [Background] Akinsola EF, Udoka PA. Parental influence on social anxiety in children and adolescents: Its assessment and management using psychodrama. Psychology. 2013; 4(3):246-53.
- [Background] Moreno TZ. To dream again (p.257). 2012; Ed.Mental Health Resources
- [Background] Ron Y. Psychodrama's Role in Alleviating Acute Distress: A Case Study of an Open Therapy Group in a Psychiatric Inpatient Ward. Front Psychol. 2018 Oct 30;9:2075. doi: 10.3389/fpsyg.2018.02075. eCollection 2018. PMID 30425674
- [Background] Croce EB. La realtà in gioco. Reale e realtà in psicodramma analitico. 2001; Rome, Italy: Borla.
- [Background] Kipper DA, Ritchie TD. The effectiveness of psychodramatic techniques: a meta-analysis. Group Dynamics: Theory, Research and Practice 2003; 7(1): 13-25.
- [Background] Qureshi AA, Awosika O, Baruffi F, Rengifo-Pardo M, Ehrlich A. Psychological Therapies in Management of Psoriatic Skin Disease: A Systematic Review. Am J Clin Dermatol. 2019 Oct;20(5):607-624. doi: 10.1007/s40257-019-00437-7. PMID 30937679
- [Background] Erbay LG, Reyhani I, Unal S, Ozcan C, Ozgocer T, Ucar C, Yildiz S. Does Psychodrama Affect Perceived Stress, Anxiety-Depression Scores and Saliva Cortisol in Patients with Depression? Psychiatry Investig. 2018 Oct;15(10):970-975. doi: 10.30773/pi.2018.08.11.2. Epub 2018 Oct 11. PMID 30301307
- [Background] Gulassa D, Amaral R, Oliveira E, Tavares H. Group therapy for excoriation disorder: Psychodrama versus support therapy. Ann Clin Psychiatry. 2019 May;31(2):84-94. PMID 31046029